CLINICAL TRIAL: NCT02903797
Title: The Relation Between Serum Irisin Hormone Level and Endometrial Hyperplasia
Brief Title: Irisin Hormone Levels in Endometrial Hyperplasia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kayseri Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Erdem Sahin, Principal Investigator, Kayseri Education and Research Hospital
Other Study IDs: 2016/466
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Endometrial Hyperplasia
Keywords: Endometrial hyperplasia; Irisin; fibronectin type III domain containing 5; FNDC5 (fibronectin type III domain containing )
MeSH Terms: conditions — Endometrial Hyperplasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Endometrial Hyperplasia: The first group was formed of the patients diagnosed endometrial hyperplasia histopathologically
- Control group: The control group was formed of the patients who were healthy women admitted to the clinic just for annual examination without any complain and symptoms

SUMMARY:
The purpose of the study is to determine serum irisin hormone levels an its relation between endometrial hyperplasia

DETAILED DESCRIPTION:
The study consisted of two groups. The first group was formed of the patients diagnosed endometrial hyperplasia histopathologically , and the controls were healthy women admitted to the clinic just for annual examination without any complain and symptoms. Patients in the 35-50 age range in both groups were included in the study. The histopathologic diagnosis of patients was established for Kayseri Education and Research Hospital Pathology clinics. Demographic parameters such as age, menopausal status, body mass index (BMI), body weight and known familial cancer story were registered.

Pregnancy, liver function disorders, cardiovascular disease, metabolic disease, diabetes, chronic kidney disease, central nerves system disease, immunosuppressive drug use, another known malignancy and excessive exercises in among one month were all exclusion criteria for the patients.

3 cc peripheral venous blood samples were taken in the patients' diagnosed endometrial hyperplasia in the course of evaluation the biopsy results and in controls during their examinations just for only once. Blood samples were centrifuged in 3200 rpm speed for 10 minutes, and stored in -80 'C until the analysis. Blood samples were evaluated on the same day after four mounts for stored first blood sample. Serum Irisin levels were evaluated with enzyme- linked immunosorbent assays kit (Catalog number: K4761-100 Biovision USA) in Kayseri Research and Education Hospital Biochemical Clinics.

ELIGIBILITY:
Inclusion Criteria:

* between 35-50 years of age
* İn endometrial hyperplasia group; patients who were diagnosed endometrial hyperplasia histopathologically

Exclusion Criteria:

* Pregnancy
* Liver function disorders
* Cardiovascular disease
* Metabolic disease
* Diabetes
* Chronic kidney disease
* Central nerves system disease
* Immunosuppressive drug use
* Another known malignancy
* Excessive exercises in among one month

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study consisted of two groups. The first group was formed of the patients diagnosed endometrial hyperplasia histopathologically, and the controls were healthy women admitted to the clinic just for annual examination without any complain and symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-01 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Serum irisin hormone levels in endometrial hyperplasia | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Erdem SAHİN, Principal Investigator — Kayseri Training and Research Hospital
Locations (1):
- Kayseri Training and Research Hospital, Kayseri, Turkey (Türkiye)